CLINICAL TRIAL: NCT04359979
Title: Treatment With Tamsulosin for Upper Eyelid Retraction Related to Thyroid Eye Disease.
Brief Title: Tamsulosin for Thyroid Lid Retraction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Oded Sagiv, Principal Investigator, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-20-7022-OS-CTIL
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Thyroid Eye Disease; Eyelid Diseases
Keywords: eyelid retraction; tamsulosin; alpha receptor antagonist
MeSH Terms: conditions — Graves Ophthalmopathy; Eyelid Diseases | interventions — Tamsulosin

STUDY DESIGN:
Intervention Model Description: off label use of an approved drug for new indication
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tamsulosin treatment (Experimental): patients will receive 0.4mg/day of Tamsulosin tablet for 3 months
  Interventions: Drug: Tamsulosin

INTERVENTIONS:
Drug: Tamsulosin — selective alpha1 receptor antagonist
  Other Names: Omnic

SUMMARY:
The purpose of this study is to examine the effect of using Tamsulosin for treatment of eyelid retraction as part of thyroid eye disease. The treatment will be offered to all thyroid patients suffering from eyelid retraction who are treated at the thyroid clinic in Sheba's Ophthalmology department. All patient will receive information about the drug Tamsulosin, the possible side effects, and the alternative treatment options for retraction.

Patients recruited will take 0.4mg/day Tamsulosin for 3 months and will have follow-ups at 1 week, 1 month and 3 months to evaluate the retraction status.

DETAILED DESCRIPTION:
Thyroid eye disease is a common autoimmune disorder caused by antibodies directed against receptors present in the thyroid cells and extra-ocular muscles and soft tissue of the orbit. The disorder is characterised by enlargement of the extra-ocular muscles, fatty and connective tissue volume.

Upper lid retraction is the most common sign of the eye disease (present in up to 92%). The causes for retraction are not fully understood. It may be related to inflammation of the Levator muscle and the Muller muscle, or related to over sympathetic activity causing overstimulation of the Muller muscle.

Upper lid retraction severity can range from very light to severe, with scleral show, eye dryness and even exposure keratopathy. Additionally it can have a very significant effect on the patient's appearance (a constant surprised look).

Treatments for lid retraction include aggressive lubrication and tarsorrhaphy if needed (sewing the eyelids together).

The Muller is a smooth muscle which elevates the upper eyelid and is sympathetically innervated (alpha receptor).

The drug Tamsulosin which is a selective alpha1 receptor antagonist is commonly used today for benign prostatic hyperplasia (relaxing the prostate muscle).

In this study we would like to test using Tamsulosin for treatment of lid retraction caused by thyroid eye disease. We hypothesise that the relaxation of the Muller muscle may have a beneficial effect on the retraction.

ELIGIBILITY:
Inclusion Criteria:

* Thyroid eye disease patients suffering from upper eyelid retraction in one or both eyes

Exclusion Criteria:

* pregnant/breastfeeding women
* previous eyelid surgery/trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
eyelid retraction | 1 week after starting tamsulosin treatment
  measuring the upper margin to reflex distance (MRD1)
eyelid retraction | 1 month after starting tamsulosin treatment
  measuring the upper margin to reflex distance (MRD1)
eyelid retraction | 3 months after starting tamsulosin treatment
  measuring the upper margin to reflex distance (MRD1)

CONTACTS AND LOCATIONS:
Overall Officials: Oded Sagiv, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yano S, Hirose M, Nakada T, Nakayama J, Matsuo K, Yamada M. Selective alpha 1A-adrenoceptor stimulation induces Mueller's smooth muscle contraction in an isolated canine upper eyelid preparation. Curr Eye Res. 2010 May;35(5):363-9. doi: 10.3109/02713680903518858. PMID 20450248
- [Background] Kikuchi-Utsumi K, Ishizaka M, Matsumura N, Nakaki T. Alpha(1A)-adrenergic control of piloerection and palpebral fissure width in rats. Auton Neurosci. 2013 Dec;179(1-2):148-50. doi: 10.1016/j.autneu.2013.04.011. Epub 2013 May 20. PMID 23701912
- [Background] Esmaeli-Gutstein B, Hewlett BR, Pashby RC, Oestreicher J, Harvey JT. Distribution of adrenergic receptor subtypes in the retractor muscles of the upper eyelid. Ophthalmic Plast Reconstr Surg. 1999 Mar;15(2):92-9. doi: 10.1097/00002341-199903000-00005. PMID 10189635